CLINICAL TRIAL: NCT05555771
Title: Determining the Effectiveness of Counterpressure Maneuvers in Pediatric Patients Presenting With Syncope to the Emergency Department
Brief Title: Paediatric Syncope in the Emergency Department
Acronym: DETECT-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Victoria Claydon (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); University of British Columbia (Other); Simon Fraser University (Other)
Responsible Party: Sponsor-Investigator, Dr. Victoria Claydon, Professor, Simon Fraser University
Organization: Simon Fraser University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-01749
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance
MeSH Terms: conditions — Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counterpressure Maneuvers (Experimental): Participants will receive standard of care treatment (behavioural intervention and avoidance measures, as indicated in "Usual Care"), alongside training in counter pressure maneuvers. Training in counterpressure maneuvers will be delivered through a handout and video that will show three maneuvers (i.e. arm-tensing, squatting, and leg-crossing) that patients enrolled in the intervention arm can perform when they begin to experience common signs and symptoms of syncope. Patients will be instructed to start with one of the maneuvers and if their symptoms do not go away, move on to a second or third maneuver if needed.
  Interventions: Behavioral: Counterpressure Maneuvers
- Usual Care (Active Comparator): Participants will receive standard of care treatment for their diagnosis of syncope. This primarily includes behavioural interventions and avoidance measures (e.g., stay hydrated, increase salt intake, avoid hot situations, avoid standing for long periods of time, engage in regular physical activity). Some patients may be prescribed medication (Midodrine, Fludrocortisone) at the discretion of their physician.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Counterpressure Maneuvers — Movements that can aid in delaying or preventing syncope by recruiting skeletal muscle pumping (via compression of major veins by contracting muscle to eject blood through cardiovascular circuit) and increased sympathetic drive (via sustaining an isometric muscle contraction). In this trial, we will be evaluating three commonly recommended maneuvers of arm tensing, squatting, and leg crossing with arm tensing. Maneuvers should be held for 1-2 minutes, or until symptoms subside.
  Other Names: Physical counter maneuvers, counter maneuvers,
  Arms: Counterpressure Maneuvers
Behavioral: Usual Care — Participants will engage in behavioural interventions and avoidance measures that are commonly recommended as a part of usual care for recurrent syncope. This primarily includes recommendations such as staying hydrated, increasing salt intake, avoiding warm temperatures, avoiding standing for long periods of time, and engaging in regular physical activity. Some patients may be prescribed medication (Midodrine, Fludrocortisone), or other assistive interventions (e.g., compression stockings) at the discretion of their physician.
  Arms: Usual Care

SUMMARY:
The investigators will assess the efficacy of clinically recommended counterpressure maneuvers (CPM) in preventing syncope for paediatric patients. Participants presenting to the emergency department (ED) will first provide written informed consent. In stage I, they will be asked to complete a brief survey documenting the presentation of their syncopal episode, and any prodromal symptoms they experienced. Participants that consent to the second stage of the study will either receive usual care (control arm) or training in counter pressure maneuvers alongside usual care (intervention arm; leg crossing, bending, arm tensing). These patients will be followed for one years time, and will be asked to complete monthly surveys detailing their syncopal and presyncopal recurrence. Medical records will be accessed over the duration of the study to identify any changes in medical diagnosis.

DETAILED DESCRIPTION:
Knowledge Gaps and Objectives The typical presentation and management for paediatric syncope is poorly understood. From research in adults, it is known that obtaining a detailed history of prodromal symptoms and the circumstance of a syncopal event is important for diagnosis, risk stratification, and determining patient prognosis. However, research in paediatric patients is lacking, with recommendations often disputed and based on a paucity of direct evidence, assuming that children will respond similarly to adults; however, this may not be the case. The investigators will (stage I) catalogue the syncopal symptoms observed in paediatric patients presenting to the emergency department (ED) with transient loss of consciousness, and (stage II) assess the efficacy of counter pressure maneuver (CPM) training in preventing recurrent syncope for paediatric patients.

Methods, Stage I; Presentation of syncope in paediatric patients Ethical approval for this study was granted by the University of British Columbia's Clinical Research Ethics Board. The investigators will recruit paediatric patients (age 7-19 years) presenting to the ED with resolved transient loss of consciousness in the last week. Research assistants will identify potential participants based on exclusion criteria, and a clinician will later gather a brief medical history and perform a screen for study eligibility. Exclusion criteria: suspected or confirmed cardiac arrhythmia diagnosis; traumatic head injury; new presentation of a seizure disorder or epilepsy; structural heart disease; hypoglycemia; physical and/or psychological disability associated with vasovagal syncope (VVS).

Consenting patients will complete a survey detailing the nature of their episodes in terms of the provocative situation, their signs and symptoms, and history of syncope or presyncope alongside a brief medical history (age, self-reported Tanner stage, age at onset of female menarche if applicable).

The primary outcome is to document the typical presentation of syncope and presyncope in paediatric patients identified as having experienced VVS. Additional outcomes include predictive factors for uncomplicated syncope in this population, including the influence of pubertal stage on the onset of paediatric syncope. Secondary outcomes include identifying the incidence of syncope, determining typical causes for syncope, and reporting on predictive factors for syncope secondary to other causes in this population. Bivariate analyses assessing possible associations between presenting prodromes and syncopal diagnoses will be conducted using either Fisher or Chi-square tests for categorical variables, and univariate multinomial models for continuous variables. These analyses will also be conducted adjusting for age and sex (either through regression or matching). The incidence and subtype of syncope presented will be calculated using an appropriate reference population. Qualitative data will be analyzed using a thematic approach, to identify trends in chosen variables based on patient responses.

Methods, Stage II; Paediatric counterpressure manoeuvres trial Stage I patients with a confirmed diagnosis of VVS from a clinician will be referred to stage II. Patients will be followed for one year while they implement either usual care for syncope (behavioural interventions and avoidance measures) or usual care alongside CPM use (leg crossing, hand grip, crouching). The primary outcome measure will be the time to syncopal reoccurrence over the 1-year follow up period, while secondary outcome measures include history of syncope in the prior 2 years, frequency of presyncopal episodes, preferred management strategies (CPM, or usual care), and barriers to implementing CPM. The predicted risk of syncopal reoccurrence will be identified using a logistic regression model with a covariate for treatment arm (CPM, standard of care). Outcomes will be compared between groups using the estimated risk ratio and risk difference. The Wald test for the log-odds coefficient from the logistic model will be used to test for treatment effect (level of 0.05). The investigators will also perform a Kaplan-Meier survival analysis (time to syncope recurrence), using a log-rank test and Cox proportional hazards analysis to compare curves. Qualitative follow-up call data will again be analyzed using a thematic approach.

ELIGIBILITY:
Inclusion Criteria:

1. Those between the ages of 6-18 years (inclusive)
2. Presenting to the ED daily 1000-2200 with resolved transient loss of consciousness that has occurred within the last week
3. Able to complete the survey in English
4. Willing and able to provide consent and assent

Exclusion Criteria:

1. Those with a known history of any of the following:

   * Suspected or confirmed cardiac arrhythmia diagnosis (e.g., Wolff-Parkinson-White, long QT)
   * Traumatic head injury
   * New presentation of seizure disorder
   * Epilepsy recurrence
   * Overdose, intoxication
   * Structural heart disease
2. Patients with hypoglycaemia and who are psychogenic with vasovagal syncope who do not present with prodromal symptoms
3. Previously enrolled in this study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with syncopal recurrence | One year, reported in monthly surveys.
  Participant experiences an episode of syncope (transient loss of consciousness and postural tone followed by a spontaneous recovery) over the course of the one year follow up.

SECONDARY OUTCOMES:
Syncopal incidence | One year
  Report on the incidence of syncope in our cohort
Documentation of typical prodromal symptoms | One year
  Link the prodromal symptoms of the different types of syncope in the pediatric population with the final diagnosis after at least one year of follow-up.
Number of patients with exercise-related syncope | One year
  Determine the diagnosis of pediatric patients who may experience syncope that is temporally associated to exercise
Number of patients with syncope secondary to other causes | One year
  Report on predictive factors for syncope secondary to other causes

CONTACTS AND LOCATIONS:
Overall Officials: Shubhayan Sanatani, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Primary Writing Committee; Sandhu RK, Raj SR, Thiruganasambandamoorthy V, Kaul P, Morillo CA, Krahn AD, Guzman JC, Sheldon RS; Secondary Writing Committee; Banijamali HS, MacIntyre C, Manlucu J, Seifer C, Sivilotti M. Canadian Cardiovascular Society Clinical Practice Update on the Assessment and Management of Syncope. Can J Cardiol. 2020 Aug;36(8):1167-1177. doi: 10.1016/j.cjca.2019.12.023. Epub 2020 Jul 2. PMID 32624296
- [Background] Malloy-Walton L, Tisma-Dupanovic S. The approach to pediatric syncope with exercise. HeartRhythm Case Rep. 2019 Oct 15;5(10):485-488. doi: 10.1016/j.hrcr.2019.04.012. eCollection 2019 Oct. No abstract available. PMID 33145167
- [Background] Sanatani S, Chau V, Fournier A, Dixon A, Blondin R, Sheldon RS. Canadian Cardiovascular Society and Canadian Pediatric Cardiology Association Position Statement on the Approach to Syncope in the Pediatric Patient. Can J Cardiol. 2017 Feb;33(2):189-198. doi: 10.1016/j.cjca.2016.09.006. Epub 2016 Oct 3. PMID 27838109
- [Background] van Dijk N, Quartieri F, Blanc JJ, Garcia-Civera R, Brignole M, Moya A, Wieling W; PC-Trial Investigators. Effectiveness of physical counterpressure maneuvers in preventing vasovagal syncope: the Physical Counterpressure Manoeuvres Trial (PC-Trial). J Am Coll Cardiol. 2006 Oct 17;48(8):1652-7. doi: 10.1016/j.jacc.2006.06.059. Epub 2006 Sep 26. PMID 17045903
- [Background] Runser LA, Gauer RL, Houser A. Syncope: Evaluation and Differential Diagnosis. Am Fam Physician. 2017 Mar 1;95(5):303-312. PMID 28290647
- [Background] Chen L, Zhang Q, Ingrid S, Chen J, Qin J, Du J. Aetiologic and clinical characteristics of syncope in Chinese children. Acta Paediatr. 2007 Oct;96(10):1505-10. doi: 10.1111/j.1651-2227.2007.00446.x. Epub 2007 Aug 20. PMID 17714543
- [Background] Anderson JB, Willis M, Lancaster H, Leonard K, Thomas C. The Evaluation and Management of Pediatric Syncope. Pediatr Neurol. 2016 Feb;55:6-13. doi: 10.1016/j.pediatrneurol.2015.10.018. Epub 2015 Nov 17. PMID 26706050
- [Background] van Wijnen VK, Gans ROB, Wieling W, Ter Maaten JC, Harms MPM. Diagnostic accuracy of evaluation of suspected syncope in the emergency department: usual practice vs. ESC guidelines. BMC Emerg Med. 2020 Aug 3;20(1):59. doi: 10.1186/s12873-020-00344-9. PMID 32746777
- [Background] Sheldon R, Rose S, Connolly S, Ritchie D, Koshman ML, Frenneaux M. Diagnostic criteria for vasovagal syncope based on a quantitative history. Eur Heart J. 2006 Feb;27(3):344-50. doi: 10.1093/eurheartj/ehi584. Epub 2005 Oct 13. PMID 16223744
- [Background] Calkins H, Shyr Y, Frumin H, Schork A, Morady F. The value of the clinical history in the differentiation of syncope due to ventricular tachycardia, atrioventricular block, and neurocardiogenic syncope. Am J Med. 1995 Apr;98(4):365-73. doi: 10.1016/S0002-9343(99)80315-5. PMID 7709949
- See also: Counterpressure maneuver training video - provided to all participants randomized to intervention arm — https://my.clevelandclinic.org/-/scassets/files/org/heart/disease-conditions/syncope/counter-pressure-techniques-1014